CLINICAL TRIAL: NCT02110992
Title: A Phase I Pilot Study of SBRT and Concurrent Docetaxel for Reirradiation of Locally Recurrent or Second Primary Squamous Cell Carcinoma of the Head and Neck
Brief Title: Safety Study of SBRT and Docetaxel for Locally Recurrent or Second Primary Squamous Cell Carcinoma of the Head and Neck
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCI-HN-13-001
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel; Radiosurgery; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel + Stereotactic Radiation (Experimental): Docetaxel 15mg/m2 IV weekly for 3 weeks. SBRT 25-40 Gy in 5 fractions given twice weekly with each treatment separated by > 48 hours.
  Interventions: Drug: Docetaxel; Radiation: Stereotactic Radiation

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 15mg/m2 IV, given days 1, 8, and 15 during SBRT
  Other Names: Taxotere; NDC 0075-8001-20
Radiation: Stereotactic Radiation — SBRT will be given over 5 fractions separated by > 48 hours. Dose will be determined based upon dose escalation schedule and will range from 25-40 Gy.
  Other Names: SBRT; Stereotactic Body Radiation; Radiation Therapy

SUMMARY:
The purpose of this research study is to test the safety of a chemotherapy drug called docetaxel and focused radiation therapy (SBRT) and see what effects (good and bad) it has on recurrent head and neck cancer that is not surgically removable.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or second primary squamous cell head and neck cancer
* Defined area of recurrence on imaging
* Previous head and neck radiation (RT) to >/= 50 Gy
* Performance status score 0-1
* Time interval from previous RT >/= 9 months
* Volume of disease appropriate for protocol treatment
* Minimum estimated survival of >/= 3 months
* Age >/= 18
* Adequate labs

Exclusion Criteria:

* Primary tumors of the salivary gland
* Original pathology report and radiation therapy records not available
* Prior spinal cord dose > 45 Gy
* Surgery or chemotherapy within 4 weeks
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years; noninvasive cancers are permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-04; Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Number of acute dose limiting toxicities | 3 months
  Acute dose limiting toxicity is defined as grade 4 or 5 toxicity measured by the Common Toxicity Criteria for Adverse Effects (CTCAE) v 4.0, including carotid arterial rupture

SECONDARY OUTCOMES:
Locoregional control | 2 years
  Time from enrollment until local failure or death (whichever comes first)
Disease-free survival | 2 years
  Time from enrollment until disease progression anywhere in the body or death (whichever comes first)
overall survival | 2 years
  Time from enrollment to death from any cause
Number of late effect dose limiting toxicities | 2 years
  Occuring > 3 months after treatment completion, including grade 4 and 5 toxicities measured by CTCAE v 4.0 involving skin, mucosa, larynx, pharynx, spinal cord, cranial nerves, and incidence of caroid blowout.

CONTACTS AND LOCATIONS:
Overall Officials: Brad Huth, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Cancer Institute, Cincinnati, Ohio, United States